CLINICAL TRIAL: NCT06384794
Title: Study of the ZyMōt Sperm Selection Method and Its Effect on Embryo Ploidy.
Acronym: ZYMOT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2211-VLC-157-MD
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Infertility, Male; Sperm Count, Low
Keywords: ZyMöt; Sperm fragmentation; Embryo development; Euploidy
MeSH Terms: conditions — Infertility, Male; Oligospermia

STUDY DESIGN:
Intervention Model Description: Multicentric, prospective, experimental study.
Who Masked: Outcomes Assessor
Masking Description: Embryologists performing IVF/ICSI are blinded to the treatment the sample has undergone. All samples are labeled with the patients Identification number. This is a unique code per patient that does not allow identification of which arm the sample belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SWIM-UP (Active Comparator): Half of the sample from the same patient will be processed by the capacitation technique routinely used in the clinic, swim-up: this is a sperm capacitation technique in which the motile spermatozoa in the seminal sample, after centrifugation and incubation, move to the top of the medium. In this way, spermatozoa with good progressive motility will remain in the supernatant.
  Interventions: Procedure: Swim-up
- ZYMOT (Experimental): Half of the semen sample will be processed through the ZyMōt® Sperm Separation Device sperm separation chip: This chip based on microfluidic properties will help us to separate and recover the semen sample with an improvement in the quality of the spermatozoa, the capacitated spermatozoa with better motility will be selected.
  Interventions: Device: Sperm capacitation through the ZyMōt®Sperm Separation Device®

INTERVENTIONS:
Device: Sperm capacitation through the ZyMōt®Sperm Separation Device® — This chip based on microfluidic properties will help us to separate and recover the semen sample with improved sperm quality. It is composed of two microwells, one initial and one final, and a porous membrane through which the sample will be filtered and the capacitated spermatozoa with better motility will be selected. Syringe 850µL of the initial seminal sample into the first well and 750µL of seminal wash medium into the second well. The device is incubated at 37°C for up to 30 minutes. During this incubation, the sample will travel by microfluidic properties from the first well through the porous membrane to the second well. This membrane will filter those spermatozoa with a higher motility. Thus, at the end of the established incubation time, the medium with the selected spermatozoa from the second well (final well) will be collected with a syringe. After this, the sample will be processed and ready for the following procedures.
  Arms: ZYMOT
Procedure: Swim-up — The swim-up is a sperm capacitation technique in which the motile spermatozoa of the seminal sample, after centrifugation and incubation, move to the upper part of the medium. In this way, spermatozoa with good progressive motility will remain in the supernatant.
  Other Names: Sperm capacitation throught swim-up technique
  Arms: SWIM-UP

SUMMARY:
It has been described that 11% of men with semen values within the normal range established by the World Health Organization (WHO) have sperm DNA fragmentation. This has been associated with a lower fertilization rate, lower embryo development and, therefore, lower reproductive success. Focusing on the study of the integrity of the male genome can provide us information to diagnose infertility in the couple. The use of conventional sperm selection methods such as swim-up or density gradients has been a great advance in the improvement of male fertility. However, these methods use centrifugation in their protocol, a procedure that has been associated with sperm DNA damage. The ZyMōt is a chip based on microfluidic properties that allows the recovery of spermatozoa with lower DNA fragmentation rate without centrifugation of the semen sample. This new sperm selection method maintains all the advantages of conventional techniques, but decreasing DNA fragmentation associates to sperm recoveries techniques eventually improving reproductive rates. This quality would be beneficial for patients with unexplained infertility, recurrent pregnancy loss or clinical varicocele, factors that have been associated with a higher index of DNA fragmentation. However up to date there is evidence-based data supporting such improvement. The main objective of the present project is to evaluate the ZyMōt as a new non-invasive sperm selection device and to see its impact on the euploidy rate, comparing it with a sperm selection technique that is routinely used in the clinic: swim-up. At the same time, the effect that this new chip may have on sperm and other reproductive variables will be analyzed clinically, and molecularly with immunohistochemical and transcriptomic analyses in order to observe the impact of SDF(sperm DNA fragmentation) at the molecular and genomic level in oocytes with low reparative potential oocytes.

ELIGIBILITY:
Inclusion Criteria:

* Couples undergoing an ICSI cycle with PGT-A (Preimplantational Genetic Test for Aneuploidy).
* Males over 18 years of age whose semen sample meets the basic conditions predetermined by the ZyMōt Multi 850µL chip.
* Fresh semen samples.
* Embryos are to be deposited in a time-lapse incubator.
* Women over 37 years of age who have obtained in follicular puncture a number of MII oocytes greater than or equal to 4.

Exclusion Criteria:

* Males with severe asthenozoospermia (<10% progressively motile spermatozoa), globozoospermia (spermatozoa with morphological alterations and lack of acrosome) and/or azoospermia (absence of spermatozoa in the ejaculate).
* Seminal samples obtained by testicular biopsy.
* Samples incubated with calcium ionophore.
* Males and females with previously known abnormal karyotype.
* Oocytes coming from the oocyte donation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
EUPLOIDY RATE | 1 YEAR
  Evaluate euploidy rate and compare it between both groups

SECONDARY OUTCOMES:
MOBILITY RATE | 1 year
  Evaluate and compare mobility between both groups
VITALITY RATE | 1 year
  Evaluate and compare vitality between both groups
DNA FRAGMENTATION RATE | 1 YEAR
  Evaluate and compare DNA fragmentation between both groups
SPERM RETRIEVAL RATE | 1 years
  Evaluate and compare sperm retrieval rate between both groups
FERTILIZATION RATE | 1 year
  Evaluate the effect of ZyMōt on the fertilization rate
USEFUL BLASTOCYS RATE | 1 year
  To evaluate number of useful blastocyst per number of MII oocyte injected and fertilized.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA JOSE DE LOS SANTOS, PhD, Principal Investigator — IVIRMA Valencia
Locations (2):
- Spain (2):
  - Ivirma Madrid, Madrid
  - Ivirma Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No